CLINICAL TRIAL: NCT00350181
Title: Sirolimus and Mycophenolate Mofetil as GVHD Prophylaxis in Myeloablative, Matched Related Donor Hematopoietic Cell Transplantation
Brief Title: Sirolimus & Mycophenolate Mofetil as GVHD Prophylaxis in Myeloablative, Matched Related Donor HCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Laura Johnston, Associate Professor of Medicine, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-06112; 97168 (Other: Stanford University); BMT184 (Other: OnCore); 6112 (Other: Stanford IRB)
Record Dates: First submitted 2006-07-05; First posted 2006-07-10 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Leukemia; Lymphoma, Non-Hodgkin; Hematologic Diseases; Acute GVHD
MeSH Terms: conditions — Leukemia; Lymphoma, Non-Hodgkin; Hematologic Diseases | interventions — Sirolimus; Mycophenolic Acid; Carmustine; Etoposide; Cyclophosphamide; Whole-Body Irradiation; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Regimen Treatment 1 (Experimental): For subjects 18-60 years old with lymphoma: (BCNU+ VP-16 +CY) BCNU 15 mg / kg (maximum dose 550 mg/m² actual body weight) on day -6. VP 60 mg / kg on day 4 and CY 100 mg / kg on day -2. Followed by Sirolimus and MMF as prophylaxis
  Interventions: Drug: Sirolimus; Drug: MMF; Drug: BCNU; Drug: VP-16; Drug: CY
- Regimen Treatment 2 (Experimental): For subjects 18-50 years old with AML, ALL or CML: (VP-16 +CY+ FBI) Patients aged 18-50 years with AML, ALL or CML: FTBI 1320 cGy delivered in 11 120 cGy fractions over 4 days on days -8 through -5. VP 60 mg / kg on day -4 and CY 60 mg / kg on day -2. Followed by Sirolimus and MMF as prophylaxis
  Interventions: Drug: Sirolimus; Drug: MMF; Drug: VP-16; Drug: CY; Drug: FTBI
- Regimen Treatment 3 (Experimental): For subjects 51-60 years with MDS, AML or ALL or 18-60 with MDS, secondary AML pr non-CML myeloproliferative disease: (BU+ VP-16 +CY) BU 1 mg/kg every 6 hours X 14 doses on days -9 through -6 with target concentration at steady state of X 800 ng / ml based on first dose pharmacokinetics. VP 60 mg / kg on day -5 and CY 45 mg / kg per day -2 days on day -3 and day -2. Followed by Sirolimus and MMF as prophylaxis
  Interventions: Drug: Sirolimus; Drug: MMF; Drug: VP-16; Drug: CY; Drug: BU

INTERVENTIONS:
Drug: Sirolimus — Immunosuppressant beginning day -3 with 12 mg oral loading dose, 4 mg/day orally for adults
  Other Names: rapamycin
Drug: MMF — Immunosuppressant given through IV on day 0 at 15 mg/kg twice daily ≥ 2hr after the completion for the donor cell infusion
  Other Names: Mycophenolate Mofetil
Drug: BCNU — 15 mg/kg, IV
  Other Names: Carmustine; BiCNU
  Arms: Regimen Treatment 1
Drug: VP-16 — 60 mg/kg, IV
  Other Names: etoposide
Drug: CY — For subjects aged 18-60 with lymphoma 100 mg/kg, IV For subjects aged with AML, ALL or CML 18-50 60 mg/kg, IV For subjects aged 51-60 with MDS, AML or ALL or patients age 18-60 with MDS, secondary AML or non-CML myeloproliferative disease 45 mg/kg
  Other Names: cyclophosphamide; cytophosphane; Endoxan
Drug: FTBI — 1320 cGy delivered in 11 120 cGy fractions over 4 day
  Other Names: total body irradiation
  Arms: Regimen Treatment 2
Drug: BU — BU 1 mg/kg every 6hr x 4 doses, IV
  Other Names: busulfan
  Arms: Regimen Treatment 3

SUMMARY:
GVHD prophylaxis of sirolimus and mycophenolate mofetil for patients undergoing matched related allogeneic transplant for acute and chronic leukemia, MDS, high risk NHL and HL

DETAILED DESCRIPTION:
To explore the novel combination of sirolimus and mycophenolate mofetil (MMF) as graft versus host disease (GVHD) prevention in HLA matched related donor blood or marrow transplantation (BMT). This study will report the toxicities associated with this drug combination and also explore possible correlations between specific blood cell types and antibody production during this therapy.

ELIGIBILITY:
Inclusion Criteria:

* Disease Categories: (one of the following)

  * AML, age 2 - 60 years beyond 2nd remission or relapsed/refractory disease
  * AML, age 51-60 years of age, in first or subsequent remission or relapsed/refractory disease
  * AML with multilineage dysplasia
  * ALL, age 2 - 60 years beyond 2nd remission or relapsed/refractory disease
  * ALL, age 51 - 60 years in first or subsequent remission or relapsed/refractory disease
  * CML Beyond 2nd chronic phase or in blast crisis
  * MDS; Includes World Health Organization classifications of refractory anemia with excess blasts-1 (RAEB-1), RAEB-2 and therapy-related MDS
  * Myeloproliferative disorders; MDS with poor long-term survival including myeloid metaplasia and myelofibrosis
  * High risk NHL in first remission
  * Relapsed or refractory NHL
  * HL beyond first remission
* Males and females of any ethnic background 2 - 60 years of age
* Karnofsky Performance Status ≥ 70% or Lansky performance status > 70% for patients < 16 years of age.
* Matched related donor identified: 6/6 HLA-A, B and DRB1
* Willingness to take oral medications during the transplantation period
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior myeloablative allogeneic or autologous HCT
* HIV infection
* Pregnant
* Lactating females
* Evidence of uncontrolled active infection
* Organ Dysfunction:
* Serum creatinine > 1.5 mg/dL or 24 hour creatinine clearance < 50 ml/min
* Direct bilirubin, ALT or AST > 2 x ULN
* In adults DLCO < 60% predicted and in children room air oxygen saturation < 92%
* In adults, left ventricular ejection fraction < 45% and in children, shortening fraction < 26%
* Fasting Cholesterol > 300 mg/dL or Triglycerides > 300 mg/dL while on lipid-lowering agents.
* Patients receiving investigational drugs unless cleared by the PI.
* Patients with prior malignancies except basal cell carcinoma or treated carcinoma in-situ.
* Cancer treated with curative intent > 5 years will be allowed.
* Cancer treated with curative intent ≤ 5 years will not be allowed with PI approval.

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2006-08; Primary Completion 2007-08 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the incidence of grade II-IV acute GVHD with sirolimus and mycophenolate mofetil GVHD prophylaxis. | D+100 post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Laura Johnston, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Johnston L, Florek M, Armstrong R, McCune JS, Arai S, Brown J, Laport G, Lowsky R, Miklos D, Shizuru J, Sheehan K, Lavori P, Negrin R. Sirolimus and mycophenolate mofetil as GVHD prophylaxis in myeloablative, matched-related donor hematopoietic cell transplantation. Bone Marrow Transplant. 2012 Apr;47(4):581-8. doi: 10.1038/bmt.2011.104. Epub 2011 May 9. PMID 21552302